CLINICAL TRIAL: NCT01697319
Title: A Phase 2, Open-label, Multinational Study to Evaluate the Efficacy and Safety of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome) Who Have Limited Ambulation
Brief Title: Efficacy and Safety Study of BMN 110 for Morquio A Syndrome Patients Who Have Limited Ambulation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR-006; 2011-005703-33 (EudraCT Number)
Record Dates: First submitted 2012-09-17; First posted 2012-10-02 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Mucopolysaccharidosis IVA; Morquio A Syndrome; MPS IVA
Keywords: Mucopolysaccharidosis IVA Type A; MPS IVA Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT; MOR-006; CPET; Limited ambulation; Grip/ Pinch
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — GALNS protein, human; Chondroitinases and Chondroitin Lyases; Galns protein, mouse; Sulfatases; Enzyme Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMN 110 at 2.0 mg/kg/week (Experimental): Weekly IV infusions of BMN 110 at 2.0 mg/kg/week over a period of approximately 4 hours per infusion for up to 144 weeks.
  Interventions: Drug: BMN 110

INTERVENTIONS:
Drug: BMN 110 — Drug will be delivered through a 4 hour (approximate) IV infusion at a dosage amount of 2.0 mg/kg/week for up to 144 weeks of treatment.
  Other Names: N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT; elosulfase alfa

SUMMARY:
The primary objective of this study is to evaluate the effect of 2.0 mg/kg/week BMN 110 in a patient population that has limited ambulation, in a period of up to 144 weeks.

DETAILED DESCRIPTION:
Effect is defined by the following key domains:

* Upper extremity function and dexterity
* Mobility

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written, signed informed consent (or their legally authorized representative) after the nature of the study has been explained and prior to performance of any research-related procedure. Patients who do not meet country and local age requirements for informed consent must be willing and able to provide written assent after the nature of the study has been explained and prior to performance of any research-related procedure.
* Has documented clinical diagnosis of MPS IVA based on clinical signs and symptoms of MPS IVA and documented reduced fibroblast or leukocyte GALNS enzyme activity or genetic testing confirming diagnosis of MPS IVA.
* Is ≥ 5 years of age.
* If sexually active, is willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at the Screening Visit and be willing to have additional pregnancy tests during the study.
* Is willing and able to perform all study procedures as physically possible.

Exclusion Criteria:

* Is able to walk farther than a specified distance as assessed by the 6MWT.
* Has previous hematopoietic stem cell transplant (HSCT).
* Has received previous treatment with BMN 110.
* Has a known hypersensitivity to any of the components of BMN 110.
* Has had major surgery within 3 months prior to study entry or is planning to have a major surgery during the first 24 weeks of the study.
* Has used any other investigational product or investigational medical device within 30 days prior to the Screening Visit or requires any investigational agent prior to completion of all scheduled study assessments.
* Is pregnant or breastfeeding at the Screening Visit or planning to become pregnant (self or partner) at any time during the study.
* Has a concurrent disease or condition, including but not limited to symptomatic cervical spine instability or severe cardiac disease or complete paralysis due to a spinal cord injury (defined as an inability to move arms and legs), that would interfere with study participation or safety as determined by the Investigator.
* Has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Decker, M.D., Study Director — BioMarin Pharmaceutical
Locations (7):
- United States (2):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
- Germany (2):
  - Universitätsklinikum Hamburg, Hamburg
  - University Medical Center Mainz, Center of Pediatric and Adolescent Medicine Villa Metabolica, Mainz
- United Kingdom (3):
  - NIHR/Wellcome Trust Birmingham CRF, Queen Elizabeth Hospital, Birmingham
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Salford Royal NHS Foundation Trust, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 110 at 2.0 mg/kg/Week: Weekly IV infusions of BMN 110 at 2.0 mg/kg/week over a period of approximately 4 hours per infusion for an initial treatment phase of 48 weeks and an extension treatment phase of up to an additional 96 weeks.
Period: Primary Phase
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Started | 16 (One subject enrolled but did not receive a single dose of study drug)
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Extension Phase
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Started | 15
Completed | 0
Not Completed | 15
Not completed — Terminated by Sponsor | 15

BASELINE CHARACTERISTICS:
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (8.38)
Age, Customized [Number; unit: participants]
  5 to 11 years | 1
  12 to 18 years | 8
  >=19 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  Other | 1
Region of Enrollment [Number; unit: participants]
  Germany | 6
  United Kingdom | 4
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Speed as Measured in Functional Dexterity Test (FDT)
Description: FDT assesses the ability to use the hand in daily tasks. The test involves turning 16 wooden pegs over as quickly as possible on a hardwood pegboard with one hand requiring a three-jaw chuck prehension pattern between the fingers and thumb within a two-minute time limit. Hand function is evaluated by how fast a patient can turn over pegs in the given time limit, i.e. speed (number of pegs/minute).
Time Frame: Up to 96 weeks
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: % of change
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Number analyzed (Participants) | 15
% of change
  Dominant Hand Wk 24 % Chg from Baseline | 1.8 (45.60)
  Dominant Hand Wk 48 % Chg from Baseline | 23.1 (53.88)
  Dominant Hand Wk 72 % Chg from Baseline | 37.2 (54.94)
  Dominant Hand Wk 96 % Chg from Baseline | 22.5 (42.21)
  Non-Dominant Hand Wk 24 % Chg from Baseline | 13.8 (32.54)
  Non-Dominant Hand Wk 48 % Chg from Baseline | 6.0 (35.78)
  Non-Dominant Hand Wk 72 % Chg from Baseline | 49.3 (126.26)
  Non-Dominant Hand Wk 96 % Chg from Baseline | -2.0 (2.83)

2. Secondary Outcome: Percent Change From Baseline in Normalized Urine Keratan Sulfate (uKS)
Description: Urinary keratan sulfate and urinary creatinine were measured through quantitative analysis. uKS is normalized to creatinine.
Time Frame: Up to 96 weeks
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: % of change
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Number analyzed (Participants) | 15
% of change
  Week 24 % Change from Baseline | -47.7 (15.40)
  Week 48 % Change from Baseline | -43.4 (24.82)
  Week 72 % Change from Baseline | -45.5 (19.67)
  Week 96 % Change from Baseline | -48.3 (24.13)

3. Primary Outcome: Change From Baseline in Strength as Assessed by Grip and Pinch Test (GPT)
Description: A grip-strength dynamometer and a pinch meter were used to measure grip strength and pinch strength. The results report change from baseline in strength for dominant and non-dominant hand in a forearm and wrist supported position.
Time Frame: Up to 96 weeks
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Number analyzed (Participants) | 15
kg
  Grip Dominant Hand Wk 24 Chg from Baseline | 0.1 (0.89)
  Grip Dominant Hand Wk 48 Chg from Baseline | -0.3 (0.90)
  Grip Dominant Hand Wk 72 Chg from Baseline | -0.1 (0.33)
  Grip Dominant Hand Wk 96 Chg from Baseline | 0.3 (0.23)
  Grip Non-Dominant Hand Wk24 Chg from Baseline | -0.0 (0.70)
  Grip Non-Dominant Hand Wk 48 Chg from Baseline | -0.1 (0.66)
  Grip Non-Dominant Hand Wk 72 Chg from Baseline | 0.1 (0.79)
  Grip Non-Dominant Hand Wk 96 Chg from Baseline | 0.4 (0.87)
  Pinch Dominant Hand Wk 24 Chg from Baseline | -0.1 (0.32)
  Pinch Dominant Hand Wk 48 Chg from Baseline | -0.0 (0.30)
  Pinch Dominant Hand Wk 72 Chg from Baseline | -0.1 (0.23)
  Pinch Dominant Hand Wk 96 Chg from Baseline | -0.6 (NA) — One observation only
  Pinch Non-Dominant Hand Wk 24 Chg from Baseline | -0.0 (0.18)
  Pinch Non-Dominant Hand Wk 48 Chg from Baseline | 0.0 (0.27)
  Pinch Non-Dominant Hand Wk 72 Chg from Baseline | -0.1 (0.31)
  Pinch Non-Dominant Hand Wk 96 Chg from Baseline | -0.3 (0.36)

4. Primary Outcome: Percent Change From Baseline in Speed as Measured in Timed 25-Foot Walk Test (25FWT)
Description: The timed 25-Foot Walk Test (25FWT) is an assessment of mobility and performance of leg function. The patient was instructed to walk a marked 25-foot course as quickly as possible in a time limit of 3 minutes and immediately walk back the same distance when reaching one end.The patient is allowed to use any ambulation method to move. The outcome measures the speed (feet / min) of moving.
Time Frame: Up to 96 weeks
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: % of change
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Number analyzed (Participants) | 15
% of change
  Wk 24 % Change from Baseline Two Attempts Combined | 95.7 (142.37)
  Wk 48 % Change from Baseline Two Attempts Combined | 53.5 (102.74)
  Wk 72 % Change from Baseline Two Attempts Combined | 48.3 (145.01)
  Wk 96 % Change from Baseline Two Attempts Combined | NA (NA) — Small sample size and zero denominators

ADVERSE EVENTS:
Time Frame: Study Period
Description: All Adverse Events
Arm/Group | BMN 110 at 2.0 mg/kg/Week
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 110 at 2.0 mg/kg/Week (N=15)
Hypersensitivity (Immune system disorders) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Central venous catheterisation (Surgical and medical procedures) | 1 (1)
Poor venous access (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 110 at 2.0 mg/kg/Week (N=15)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Otorrhoea (Ear and labyrinth disorders) | 1 (2)
Corneal opacity (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eyelid cyst (Eye disorders) | 1 (1)
Eyelid pain (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (7)
Abdominal pain upper (Gastrointestinal disorders) | 6 (12)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (28)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (19)
Vomiting (Gastrointestinal disorders) | 6 (29)
Catheter site pain (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Device occlusion (General disorders) | 2 (2)
Extravasation (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Feeling cold (General disorders) | 2 (2)
Influenza like illness (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (2)
Infusion site pain (General disorders) | 1 (3)
Infusion site reaction (General disorders) | 1 (5)
Injection site pain (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (2)
Medical device pain (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (5)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 4 (5)
Pyrexia (General disorders) | 9 (26)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Anaphylactoid reaction (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Reaction to colouring (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (3)
Bronchitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (2)
Ear infection (Infections and infestations) | 2 (5)
Eye infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4)
Nasopharyngitis (Infections and infestations) | 9 (19)
Otitis externa fungal (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (2)
Periodontitis (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 3 (4)
Skin candida (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (14)
Urinary tract infection (Infections and infestations) | 1 (6)
Viral infection (Infections and infestations) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (2)
Electrocardiogram PR prolongation (Investigations) | 1 (1)
QRS axis abnormal (Investigations) | 2 (2)
Weight increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (16)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Clonus (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 4 (10)
Headache (Nervous system disorders) | 11 (42)
Hypoaesthesia (Nervous system disorders) | 1 (3)
Lethargy (Nervous system disorders) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (14)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (6)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Poor venous access (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days